CLINICAL TRIAL: NCT01225159
Title: Safety and Efficacy of Tight Glycaemic Control During Cardiac Surgery
Brief Title: Tight Glycaemic Control During Cardiac Surgery
Acronym: TGC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Hypoglycaemia is significantly higher in TGC
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Panthila Rujirojindakul, Assistant Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SUB.EC 51-1008-08-1-1
Record Dates: First submitted 2010-07-29; First posted 2010-10-20 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Nosocomial Infection; External Causes of Morbidity and Mortality; Hypoglycemia
Keywords: tight glycemic control; cardiac surgery
MeSH Terms: conditions — Cross Infection; Hypoglycemia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tight glycaemic control (TGC) (Experimental): TGC used hyperinsulinaemic normoglycaemic clamp with modified glucose-insulin-potassium to control blood sugar. The insulin (HumulinTM R, Lilly pharma, Germany) was diluted with normal saline to the concentration 1 IU. mL-1 and was infused continuously throughout the operations at a fixed rate of 0.3 IU. kg-1.h-1 but the maximal rate was 20 IU/ h. A separate mixture of glucose 25% (A.N.B Laboratories, Thailand) 50 mL, potassium chloride (Nida pharma, Thailand) 20 mEq and magnesium sulfate (Atlantic, Thailand) 2 gm was infused at 0.75 mL.kg-1.h-1 and was adjusted to maintain blood glucose levels 80-150 mg/dL.
  Interventions: Drug: TGC
- Conventional glycaemic control (Control) (Placebo Comparator): Conventional glycaemic control aims to control blood sugar less than 250 mg%. Insulin was given bolusly if the blood sugar more than 250 mg%.
  Interventions: Drug: Conventional glycaemic control

INTERVENTIONS:
Drug: TGC — TGC used hyperinsulinaemic normoglycaemic clamp with modified glucose-insulin-potassium to control blood sugar. The insulin (HumulinTM R, Lilly pharma, Germany) was diluted with normal saline to the concentration 1 IU. mL-1 and was infused continuously throughout the operations at a fixed rate of 0.3 IU. kg-1.h-1 but the maximal rate was 20 IU/ h. A separate mixture of glucose 25% (A.N.B Laboratories, Thailand) 50 mL, potassium chloride (Nida pharma, Thailand) 20 mEq and magnesium sulfate (Atlantic, Thailand) 2 gm was infused at 0.75 mL.kg-1.h-1 and was adjusted to maintain blood glucose levels 80-150 mg/dL.
  Other Names: intensive glycaemic control
  Arms: Tight glycaemic control (TGC)
Drug: Conventional glycaemic control — Conventional glycaemic control aims to control blood sugar less than 250 mg%. Insulin was given bolusly if the blood sugar more than 250 mg%.
  Other Names: Control group
  Arms: Conventional glycaemic control (Control)

SUMMARY:
To determine whether intraoperative tight glycaemic control can reduce postoperative infection, morbidity and mortality

DETAILED DESCRIPTION:
Hyperglycaemia develops frequently in patients undergoing cardiac surgery, especially following cardiopulmonary bypass (CPB). Recent evidence suggests that acute hyperglycaemia adversely affects immune function, wound healing and cardiovascular function.

ELIGIBILITY:
Inclusion Criteria:

* age > 15 years
* cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* active infection
* insulin allergy
* off-pump cardiopulmonary bypass procedures

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panthila Rujirojindakul, M.D., Principal Investigator — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Faculty of Medicine, PSU, Hat Yai, Changwat Songkhla, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Tight Glycaemic Control (TGC): Allocated to intensive group (n = 100)
  * Received allocated intervention (n = 99)
  * Did not receive allocated intervention: change operation (n = 1)
- Conventional Glycaemic Control (Control): Allocated to control group (n = 100)
  • Received allocated intervention (n = 100)
Period: Overall Study
Arm/Group | Tight Glycaemic Control (TGC) | Conventional Glycaemic Control (Control)
Started | 100 | 100
Completed | 99 | 100
Not Completed | 1 | 0
Not completed — Change operation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline and clinical characteristics of the study patients did not significantly differ between the two groups. There were 18 diabetic patients in the intensive group and 17 diabetic patients in the control group, and there was no difference in terms of the diabetic treatment given (P = 0.77).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tight Glycaemic Control (TGC) | Conventional Glycaemic Control (Control) | Total
Number analyzed (Participants) | 99 | 100 | 199
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [38.0 to 63.5] | 54 [45.0 to 65.2] | 54 [41.5 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 55 | 57 | 112
Mean body mass index (SD), kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 22.7 (3.9) | 23.3 (4.4) | 22.8 (4.1)
Smoking status [Number; unit: participants]
  Current | 21 | 11 | 32
  Former | 28 | 32 | 60
  Never | 48 | 53 | 101
  No data | 2 | 4 | 6
New York Heart Association (NYHA) class [Number; unit: participants] — Class I: Cardiac disease, but no symptoms and no limitation in ordinary physical activity, Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity, Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, Class IV: Severe limitations. Experiences symptoms even while at rest.
  participants
    1 | 8 | 5 | 13
    2 | 55 | 65 | 120
    3 | 32 | 25 | 57
    4 | 4 | 5 | 9
American Society of Anesthesiologists (ASA) class [Number; unit: participants] — ASA classification defined according to American Society of Anesthesiologists that divided into 4 classes:
  ASA class 1: healthy patient ASA class 2: mild systemic disease ASA class 3: uncontrolled systemic disease ASA class 4: incapacitated patient ASA class 5: moribund
  participants
    3 | 86 | 87 | 173
    4 | 12 | 10 | 22
    5 | 1 | 3 | 4
Operation [Number; unit: participants]
  Valve replacement / repairment | 39 | 43 | 82
  Coronary artery bypass graft | 37 | 37 | 74
  Closure of septal defects | 10 | 5 | 15
  Bentall's operation | 1 | 1 | 2
  Aneurysmectomy of thoracic aortic aneurysm (TAA) | 0 | 3 | 3
  More than 1 operation | 7 | 8 | 15
  Others | 5 | 3 | 8
Case status [Number; unit: participants]
  Elective | 76 | 72 | 148
  Emergency | 23 | 28 | 51
Underlying disease:DM [Number; unit: participants]
  Yes | 18 | 17 | 35
  No | 81 | 83 | 164

OUTCOME MEASURES:

1. Primary Outcome: Nosocomial Infection
Description: Infection rate referred to the rate of nosocomial infection, including pneumonia, central line infection, surgical wound infection, deep sternal wound infection, urinary tract infection, and sepsis. Infections were defined according to the Centers for Disease Control and Prevention (CDC) definitions, occurring within 30 days postoperative cardiac surgery.
Time Frame: within the first 30 day after surgery
Measure: Number; unit: participants
Groups:
- Tight Glycaemic Control (TGC): Allocated to control group (n = 100)
  * Received allocated intervention (n = 99)
  * Did not receive allocated intervention: change operation (n = 1)
- Conventional Glycaemic Control (Control): Allocated to intensive group (n = 100)
  • Received allocated intervention (n = 100)
Arm/Group | Tight Glycaemic Control (TGC) | Conventional Glycaemic Control (Control)
Number analyzed (Participants) | 99 | 100
participants | 17 | 13

2. Secondary Outcome: Morbidities and All Causes Mortality
Description: morbidities defined as hypoglycaemia (blood sugar less than 60 mg/dL), Stroke (focal neurological deficit confirmed with CT or MRI), acute renal failure (rising of creatinine)
Time Frame: within the first 30 days after surgery
Measure: Number; unit: participants
Arm/Group | Tight Glycaemic Control (TGC) | Conventional Glycaemic Control (Control)
Number analyzed (Participants) | 99 | 100
participants
  Hypoglycemia | 23 | 3
  Stroke | 6 | 3
  New atrial fibrillation | 17 | 21
  Acute kidney injury | 5 | 6
  Cardiac arrest | 3 | 1
  Death | 6 | 8

ADVERSE EVENTS:
Time Frame: 30 days postoperative
Arm/Group | Tight Glycaemic Control (TGC) | Conventional Glycaemic Control (Control)
Serious Adverse Events (participants affected / at risk) | 23/99 | 3/100
Other Adverse Events (participants affected / at risk) | 17/99 | 13/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tight Glycaemic Control (TGC) (N=99) | Conventional Glycaemic Control (Control) (N=100)
Hypoglycemia (Endocrine disorders) | 23 | 3 — Hypoglycemia was defined as blood glucose < 60 mg/dl ( 3.3 mmol / l).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tight Glycaemic Control (TGC) (N=99) | Conventional Glycaemic Control (Control) (N=100)
Infection rate (Infections and infestations) | 17 (17) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes